CLINICAL TRIAL: NCT05451095
Title: A Randomized, Placebo Controlled, Double-blind, Double-dummy, Three-way Crossover Trial to Investigate the Effect of Two Doses of BI 474121 on Ketamine Induced Cognitive Deficits in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test Whether BI 474121 Can Reverse the Memory Problems Caused by Ketamine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Termination of project
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1411-0003
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Healthy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment sequence T1-T2-R (Experimental): T1: Lower dose of BI 474121 and higher dose of placebo followed by intravenous ketamine infusion T2: Higher dose of BI 474121 and lower dose of placebo followed by intravenous ketamine infusion R: Lower dose of placebo and higher dose of placebo followed by intravenous ketamine infusion
  Interventions: Drug: BI 474121; Drug: Placebo; Drug: Ketamine hydrochloride
- Treatment sequence T2-T1-R (Experimental)
  Interventions: Drug: BI 474121; Drug: Placebo; Drug: Ketamine hydrochloride
- Treatment sequence T1-R-T2 (Experimental)
  Interventions: Drug: BI 474121; Drug: Placebo; Drug: Ketamine hydrochloride
- Treatment sequence T2-R-T1 (Experimental)
  Interventions: Drug: BI 474121; Drug: Placebo; Drug: Ketamine hydrochloride
- Treatment sequence R-T1-T2 (Experimental)
  Interventions: Drug: BI 474121; Drug: Placebo; Drug: Ketamine hydrochloride
- Treatment sequence R-T2-T1 (Experimental)
  Interventions: Drug: BI 474121; Drug: Placebo; Drug: Ketamine hydrochloride

INTERVENTIONS:
Drug: BI 474121 — BI 474121
Drug: Placebo — Placebo
Drug: Ketamine hydrochloride — Ketamine hydrochloride

SUMMARY:
To investigate the effect of BI 474121 compared to placebo on ketamine-induced cognitive deficits to predict efficacy in patients with cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 32 kg/m2 (inclusive)
* Signed and dated written informed consent(s) prior to admission to the study, in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* If men who are able to father a child, are willing to participate, they have to use an adequate form of effective contraception for the duration of study participation and for at least 30 days after treatment has ended

Exclusion Criteria:

* Any finding in the medical examination (including ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm evaluated as clinically significant by Investigators
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* History of diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-07 (Estimated); Primary Completion 2023-06-05 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Difference between the total number of errors adjusted for stages that subjects did not complete in the paired associate learning test (PALTEA28), post-ketamine minus the PALTEA28 pre-ketamine | up to 22 days

SECONDARY OUTCOMES:
Difference between the between errors in the spatial working memory test (SWMBE468), post-ketamine minus the SWMBE468 pre-ketamine | up to 22 days
Difference between the Rapid Visual Information Processing test A' (RVPA), post-ketamine minus the RVPA pre-ketamine | up to 22 days

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com